CLINICAL TRIAL: NCT07286890
Title: A Real-World Post-Market Clinical Follow-Up Study to Evaluate the Safety and Performance of Getinge's Beating Heart Product Family in Patients Undergoing Beating Heart Coronary Artery Bypass Graft Surgery
Brief Title: Getinge's Beating Heart Product Family Post-Market Clinical Follow-up (PMCF) Study
Status: Not yet recruiting | Type: Observational
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MCV00110458
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Off Pump Coronary Artery Bypass Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Getinge Beating heart study devices group
  Interventions: Device: Vacuum Stabilizer System; Device: Vacuum Positioner System; Device: Blower/Mister; Device: Proximal Seal System

INTERVENTIONS:
Device: Vacuum Stabilizer System — Isolates and provides local immobilization of the target vessel while performing the distal anastomosis on a beating heart.
Device: Vacuum Positioner System — Positions the heart and exposes the coronary artery(ies) when performing the distal anastomosis on a beating heart.
Device: Blower/Mister — Reduces blood in the operative field to improve visibility while performing an anastomosis on a beating heart.
Device: Proximal Seal System — Proximal anastomotic seal technology allows for clampless hemostasis during proximal anastomosis when performing Coronary Artery Bypass Graft (CABG) procedures.

SUMMARY:
This observational study aims to collect data on the performance and safety of Getinge's Beating Heart products used during open-heart coronary artery bypass graft surgery. The surgery and the use of the study devices will be done according to the standard of care. Participants will not be required to undergo any study-specific procedures, and information will be collected only until hospital discharge following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 22 years of age
* Patient (or a legally authorized representative) is willing and able to provide signed informed consent, if required
* Undergoing planned beating heart coronary artery bypass graft procedure with/without left atrial appendage closure, where the use of at least one Getinge's Beating Heart study product is anticipated.

Exclusion Criteria:

* Patients undergoing heart valve surgery
* Patients who undergo either planned or unplanned conversion to on pump with arrested heart where Getinge's Beating Heart product(s) have not been used.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing beating heart coronary artery bypass surgery where 1 or more Beating Heart study products are used according to the device labeling.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related adverse events | Time period from procedure through study completion, an average of 7 days
  Incidence of device-related adverse events for each subject
Incidence of device-related serious adverse events | Time period from procedure through study completion, an average of 7 days
  Incidence of device-related serious adverse events experienced by subjects
Incidence of technical success | Perioperative/Periprocedural
  Incidence of technical success, based on the number of patients who have documented successful use and performance of the study device(s) when used as intended, out of the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bulger, Study Director — Getinge

IPD SHARING:
Plan to Share IPD: No